CLINICAL TRIAL: NCT01561131
Title: The Effect of Protein and Calcium on Weight Change and Blood Lipid Profile
Acronym: PROKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Arla Foods (Industry); Nupo A/S, Denmark (Unknown)
Responsible Party: Principal Investigator, Arne Astrup, Prof., MD, Head of Department, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B288
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Prevention of Obesity
Keywords: Obesity; Protein intake; Calcium intake; Weight loss; Weight maintenance; Blood lipid profile; Diet induced thermogenesis
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Whey Proteins; Calcium; Soybean Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Whey protein supplement (Active Comparator): Whey protein
  Interventions: Dietary Supplement: Whey protein
- Whey protein enriched with calcium supplement (Active Comparator): Whey protein enriched with calcium
  Interventions: Dietary Supplement: Whey protein enriched with calcium
- Soy protein supplement (Active Comparator): Soy protein
  Interventions: Dietary Supplement: Soy protein
- Control supplement (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Whey protein — 45g protein/d; Dosage 3x15g protein daily
  Arms: Whey protein supplement
Dietary Supplement: Whey protein enriched with calcium — 45g protein/d + 1000mg calcium/d; dosage: 15g protein + 333mg calcium x 3 daily
  Arms: Whey protein enriched with calcium supplement
Dietary Supplement: Soy protein — 45g soy protein/d; dosage 15g soy protein x 3 daily
  Arms: Soy protein supplement
Dietary Supplement: Maltodextrin — 48g carbohydrate/d; dosage: 16g carbohydrate x 3 daily
  Arms: Control supplement

SUMMARY:
The primary aim is to examine the effect of a high protein intake (from soy or whey protein) on weightmaintenance after weight loss in a group of predisposed (severe) obese persons. Furthermore, to examine short-term and long-term effect of a high protein intake on appetite regulation and diet induced thermogenese (DIT). Finally to examine the effect of calcium on weightmaintence, bloodlipid profilen, appetite regulation and DIT.

The study is a parallel RCT with a weight loss (WL) period (8 weeks on very low calorie diet) and a weightmaintence (WM) period (24 weeks daily intake of supplement). 200 overweight/obese subjects will be enrolled into the study and randomized to placebo (maltodextrin), soy protein, whey protein or calcium enriched whey protein supplement. At baseline (week 0), after the WL period (week 8) and after WM period (week 24) body weight and composition will be measured and blood samples will be collected. Meal test will be performed at week 0 and 24 (examining both appetite regulation and DIT). Urine and feces will be collected three times during the study. Subjects will receive dietary counseling (in groups) regularly during the study and body weight will be measured at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women can be included
* All ethnic groups can be included
* Age: 18≤age≤60
* BMI: 28≤BMI≤40

Exclusion Criteria:

* smoking
* use of cholesterol-lowering medications or other medications considered to be of importance for participation in the trial
* use of special diets (eg. Atkins, vegetarian) within 2 months before the start of the project.
* elite athletes or if subjecct is planning to become elite athlete (e.g. Planning major changes in physical activity during the experiment).

  * blood donation within the last 3 months before the commencement of the trial
  * weight change> 3 kg within 2 months before the start of the project
  * sagital height of 32 cm
  * pregnant or nursing women or women planning to become pregnant within the next 12 months.
  * surgically treated obesity
  * participation in other clinical trials within the last 3 months
  * if consuming medicine daily, consumption of prescription medicine needs to have been stable through at least the last 3 months and is expected to remain so throughout the whole study. However, a subject cannot be included if the treatment includes medicine that is a systemic treatment that is considered to be of importance for participation in the project.
  * alcohol or drug use (based on clinical judgment)
  * subjects who are unable to give an informed consent.
  * chronic systemic infectious or inflammatory disorders
  * chronic endocrine disorders
  * inadequate nutrient uptake, or chronic gastrointestinal or liver diseases (apart from irritable bowel disorder)
  * cardiovascular disease, recognized heart failure or brain disease
  * cancer within the past 10 years
  * subject who is judged unable to participate in an LCD (low calorie diet) in an 8 week period
  * known allergy to para-aminobenzoic acid (PABA)
  * subjects who are in a general physical and/or mental condition,where the researcher assesses that the subject does not conform with the general aim of the study.
  * subjects with a hemoglobin value below 7 mol / L. Those with a hemoglobin value below 8 mol / L (measured at screening) cannot volunteer for the meal test during hood measurements, but may be included in the main study.

When starting on a weight maintenance period:

• persons during weight loss period, loss of <8% of their initial body weight

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Difference in body weight and composition during the weight maintenance period | 24 weeks

SECONDARY OUTCOMES:
Difference in fasting blood lipid profile during the weight maintenance period. | 24 weeks
Difference in fasting insulin, glucose, C-peptide, glucagon, insulin-like growth factor 1 (IGF-1), ionized calcium, parathyroideahormone (PTH), and angiopoietin-like protein 4 (Angpt14) during the weight maintenance period. | 24 weeks
Difference in resting blood pressure and pulse during the weight maintenance period. | 24 weeks
Difference in intestinal flora during the weight maintenance period. | 24 weeks
Nutrigenomics (NMR) analysis. | 24 weeks
Difference in energy intake (EI) and macronutrient intake from the diet during the weight maintenance period. | 24 weeks
Difference in acute- and long-term effet on diet induced thermogenesis and substrate oxidation. | 24 weeks.
Difference in acute- and long-term effect on postprandial appetite regulation (measured via VAS, appetite regulating hormones and energy intake) | 24 weeks
Difference in acute- and long-term effect on postprandial response in insulin, glucose, C-peptide, and glucagon. | 24 weeks
Difference in appetite regulating hormones (ghrelin, glucagon-like peptide-1 (GLP-1), peptide YY (PYY), and cholecystokinin (CCK)) during weight maintenance period. | 24 weeks
Change in body weight and composition during the weight loss period | 8 weeks
Change in blood lipid profile during the weight loss period | 8 weeks
Change in fasting insulin, glucose ect. during the weight loss period | 8 weeks
Change in intestinal flora during the weight loss period. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Prof., MD, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, University of Copenhagen, Frederiksberg, Copenhagen, Denmark

REFERENCES:
- [Derived] Geiker NRW, Veller M, Kjoelbaek L, Jakobsen J, Ritz C, Raben A, Astrup A, Lorenzen JK, Larsen LH, Bugel S. Effect of low energy diet for eight weeks to adults with overweight or obesity on folate, retinol, vitamin B12, D and E status and the degree of inflammation: a post hoc analysis of a randomized intervention trial. Nutr Metab (Lond). 2018 Apr 10;15:24. doi: 10.1186/s12986-018-0263-1. eCollection 2018. PMID 29643928
- [Derived] Kjolbaek L, Sorensen LB, Sondertoft NB, Rasmussen CK, Lorenzen JK, Serena A, Astrup A, Larsen LH. Protein supplements after weight loss do not improve weight maintenance compared with recommended dietary protein intake despite beneficial effects on appetite sensation and energy expenditure: a randomized, controlled, double-blinded trial. Am J Clin Nutr. 2017 Aug;106(2):684-697. doi: 10.3945/ajcn.115.129528. Epub 2017 Jul 5. PMID 28679554